CLINICAL TRIAL: NCT01482169
Title: Efficacy of Intravenous Regadenoson Versus Intravenous Adenoscan® for Fractional Flow Reserve Measurements
Brief Title: Intravenous Regadenoson Versus Intravenous Adenoscan® for Fractional Flow Reserve (FFR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Bober, M.D., Director of Nuclear Cardiology, Ochsner Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10012012
Record Dates: First submitted 2011-11-15; First posted 2011-11-30 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Left heart catheterization; Fractional flow reserve; Adenoscan®; Regadenoson
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adenoscan (Active Comparator): Subjects will have the FFR Measurement with IV Adenoscan®
  Interventions: Drug: FFR Measurement with IV Adenoscan® then with Regadenoson
- Regadenoson (Experimental): Subjects will have the FFR Measurement with IV Regadenoson
  Interventions: Drug: FFR Measurement with IV Adenoscan® then with Regadenoson

INTERVENTIONS:
Drug: FFR Measurement with IV Adenoscan® then with Regadenoson — Testing will be completed during a Left Heart Catheterization (LHC). The first 48 eligible patients enrolled will receive an initial infusion of IV Adenoscan® through a peripheral vein at 140 mcg/kg/min. FFR measurements will be obtained utilizing a coronary pressure guide wire once peak hyperemia has been achieved. It takes about 84 seconds to reach peak hyperemia with Adenoscan®. Subsequently, these subjects will receive a dose of regadenoson at 0.4 mg through the same peripheral access site. FFR measurements will be obtained once peak hyperemia is achieved, which takes less than 30 seconds with regadenoson. Patients who react to either medication will be supported conservatively under close scrutiny.
  Other Names: Adenoscan® vs Regadenoson

SUMMARY:
The purpose of this study is to demonstrate that intravenous regadenoson is equivalent to intravenous Adenoscan® for the physiological assessment of intermediate coronary lesions.

DETAILED DESCRIPTION:
This is a prospective open label, single center pilot trial that will evaluate regadenoson compared to Adenoscan® to be given IV in the assessment of Fractional Flow Reserve. Forty eight subjects will be enrolled and get Adenoscan® administered via IV followed by Regadenoson IV.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective left heart catheterization
* Age ≥ 18 years (female not of child bearing potential)
* Able to provide written informed consent

Exclusion Criteria:

* Contraindications to administration of either Adenoscan® or Regadenoson
* High degree AV block, sick sinus syndrome without a functioning pacemaker
* Symptomatic bradycardia
* Recent STEMI (< 5 days)
* Recent NSTEMI (<5 days) if the peak CK is > 1000 IU
* Dipyridamole use within 24 hours
* Adenoscan® is contraindicated (hypersensitivity to Adenoscan®, Regadenoson, or aminophylline
* Known severe bronchoconstrictive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bober, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adenoscan + Regadenoson: Subjects will have the FFR Measurement with IV Adenoscan® then with Regadenoson
  FFR Measurement with IV Adenoscan® then with Regadenoson: Testing will be completed during a Left Heart Catheterization (LHC). The first 48 eligible patients enrolled will receive an initial infusion of IV Adenoscan® through a peripheral vein at 140 mcg/kg/min. FFR measurements will be obtained utilizing a coronary pressure guide wire once peak hyperemia has been achieved. It takes about 84 seconds to reach peak hyperemia with Adenoscan®. Subsequently, these subjects will receive a dose of regadenoson at 0.4 mg through the same peripheral access site. FFR measurements will be obtained once peak hyperemia is achieved, which takes less than 30 seconds with regadenoson. Patients who react to either medication will be supported conservatively under close scrutiny.
Period: Overall Study
Arm/Group | Adenoscan + Regadenoson
Started | 48
Completed | 46
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Adenoscan + Regadenoson
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 61.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Comparing Measurement of Fractional Flow Reserve (FFR)
Description: For the first measurement of FFR, the subject will receive Adenoscan® by IV infusion. Then the FFR measurements will be taken. When vital signs have returned to normal, after two minutes the line will be flushed with saline. The subject will then receive Regadenoson by IV infusion and repeat FFR measurements will be recorded. The subject will be administered aminophylline and the time duration it takes to return to baseline hemodynamic will be recorded.
Time Frame: DAY 1
Measure: Mean (Standard Deviation); unit: FFR
Groups:
- Adenoscan: Subjects will have the FFR Measurement with IV Adenoscan®
  FFR Measurement with IV Adenoscan®: Testing will be completed during a Left Heart Catheterization (LHC). The first 48 eligible patients enrolled will receive an initial infusion of IV Adenoscan® through a peripheral vein at 140 mcg/kg/min. FFR measurements will be obtained utilizing a coronary pressure guide wire once peak hyperemia has been achieved. It takes about 84 seconds to reach peak hyperemia with Adenoscan®.
- Regadenoson: Subjects will have the FFR Measurement with IV Regadenson
  FFR Measurement with IV Regadenson: Testing will be completed during a Left Heart Catheterization (LHC). The first 48 eligible patients enrolled will receive IV Regadenson through a peripheral vein. FFR measurements will be obtained utilizing a coronary pressure guide wire once peak hyperemia has been achieved.
Arm/Group | Adenoscan | Regadenoson
Number analyzed (Participants) | 46 | 46
FFR | .83 (0.082) | .84 (0.084)

2. Secondary Outcome: Duration to Baseline Hyperemia After Aminophylline Injection
Description: In the regadenoson arm, the duration to baseline hyperemia after aminophylline Injection
Time Frame: seconds
Population: Of the 48 patients enrolled, 7 of the patients did not have measurements for the secondary outcome.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Duration to Baseline Hyperemia After Aminophylline Administrat: After subjects have the FFR measurement with Regadenoson, they will be administered aminophylline 150mg IV and the time duration to reach baseline hyperemia will be recorded.
Arm/Group | Duration to Baseline Hyperemia After Aminophylline Administrat
Number analyzed (Participants) | 41
seconds | 112 (72)

ADVERSE EVENTS:
Time Frame: Subjects were monitored during and post-procedure until discharge from the procedure. This duration was less than 24 hours for each participant.
Description: Definitions do not differ.
Groups:
- Regadenson: Subjects will have the FFR Measurement with IV Regadenson
  FFR Measurement with IV Regadenson: Testing will be completed during a Left Heart Catheterization (LHC). The first 48 eligible patients enrolled will receive IV Regadenson through a peripheral vein. FFR measurements will be obtained utilizing a coronary pressure guide wire once peak hyperemia has been achieved.
Arm/Group | Adenoscan | Regadenson
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes